CLINICAL TRIAL: NCT03262584
Title: Evaluation of NGS for Detection and Follow-up of Fungal Pathogens in Immunocompromised Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Karius, Inc. (Industry)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: KDP-001
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Invasive Fungal Disease; Fever and Neutropenia; Invasive Fungal Infections; Immunocompromised
MeSH Terms: conditions — Invasive Fungal Infections; Fever; Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Sponsor hypothesize that Next-generation Sequencing (NGS) can identify fungal pathogens, is more accurate than other noninvasive options and can report fungal genomic load.

DETAILED DESCRIPTION:
The Sponsor aims to describe the incidence of positivity for fungal specific pathogens on NGS analysis in a high-risk immunocompromised pediatric population.

Secondarily, the Sponsor will correlate results of the NGS analysis to other approved fungal tests if performed at the discretion of the treating provider (e.g. blood culture results, radiographic findings, biopsy results, bronchoalveolar lavage findings, galactomannan results or b-D-glucan (BG) results as evaluated via FDA-approved "Fungitell" assay). The Sponsor will use these other fungal tests, in addition to clinical criterion, to classify subjects as having possible, probable and proven IFD according to established criteria, and compare these categories against results from NGS analysis.

Lastly, to quantitatively evaluate follow-up test results to determine fungal DNA genomic load in subjects with positive results.

ELIGIBILITY:
Inclusion Criteria:

* Prolonged FN (≥96 hours) despite broad-spectrum antibiotic therapy with anticipated delayed neutrophil recovery
* Any findings that trigger the primary team to consider new fungal infection in a given inpatient, such as abnormal imaging results, recrudescent fevers in the setting of neutropenia or characteristic skin rashes

Exclusion Criteria:

-Those without concern for fungal infection or those currently being treated for a presumed or documented fungal infection will not be recruited for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric patients treated at Ann & Robert H. Lurie Children's Hospital of Chicago on the hematology, oncology, neuro-oncology and stem cell transplant unit
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Incidence of positivity for fungal specific pathogens on NGS analysis | 7 months
  We aim to describe the incidence of positivity for fungal specific pathogens on NGS analysis in a high-risk immunocompromised pediatric population.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Armstrong, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States